CLINICAL TRIAL: NCT01663597
Title: Optical Biometry and Spherical Aberration in Ametropic and Emmetropic Eyes
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. Doz. Dr., Medical University of Vienna
Other Study IDs: OPHTH-240512
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Refractive Errors; Axial Length, Eye; Corneal Wavefront Aberration
MeSH Terms: conditions — Refractive Errors; Corneal Wavefront Aberration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Cohort 1: 40 subjects with high grarde myopia ranging from -10 diopters to -4.01 diopters
- Cohort 2: 40 subjects with moderate myopia ranging from -4 diopters to -1.01 diopter
- Cohort 3: 40 subjects with emmetropia, -1 diopter to +1 diopter
- Cohort 4: 40 subjects with hyperopia, +1.01 diopter and more

SUMMARY:
Aberrations play a significant role in the visual process and can be divided in lower-order and higher-order aberrations. The former can be measured using the commercially available IOL Master (Carl Zeiss Meditec AG, Germany) and have profound influence on visual acuity. Higher-order aberrations do not significantly influence visual acuity but affect the quality of vision and can cause halos, double vision, and night vision disturbances.

Background Cataract surgery has become a routine procedure in the developed countries. During this surgery, a foldable intraocular lens is usually inserted into the capsular bag. However, these lenses do not account for individual optical biometry data or aberrations. Therefore, it is important to provide data for ametropic and emmetropic eyes as this information might improve future intraocular lens design and lead to individually adapted lenses for yielding optimal visual acuity and quality results.

The aim of the present study is to clarify the correlation between refractive errors/axial eye length and spherical aberrations of the cornea.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged between 40 and 60 years
* normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* normal ophthalmic findings unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* presence of any corneal or retinal disease
* Dry eye syndrome
* high astigmatism (>1 diopter)
* history of refractive surgery
* abuse of alcoholic beverages
* participation in a clinical trial in the 3 weeks preceding the study
* symptoms of a clinically relevant illness in the 3 weeks before the study day
* pregnancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants will be selected by the Department of Clinical Pharmacology
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Axial eye length | 1 day

SECONDARY OUTCOMES:
Refractive error | 1 day
Corneal radius | 1 day
Pupil diameter | 1 day
Anterior chamber depth | 1 day
Anterior corneal topography | 1 day
Corneal thickness map | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria